CLINICAL TRIAL: NCT04878237
Title: Mapping the Kinetics of Cytokine Responses to Mechanical Stimulation of the Nose in Asthmatic, Allergic and Non-Allergic Subjects - A Pilot Study
Brief Title: Kinetics of Nasal Cytokine Responses to Mechanical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sven Schneider, MD, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MUViennaAstra2021
Record Dates: First submitted 2021-04-02; First posted 2021-05-07 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis Due to Grass Pollen; Allergic Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non Allergic Patients (Placebo Comparator)
  Interventions: Other: Nasal Secretion Sampling
- Allergic Asthma Patients (Active Comparator): Allergy to Grass Pollen
  Interventions: Other: Nasal Secretion Sampling
- Allergic Rhinitis Patients (Active Comparator): Allergy to Grass Pollen
  Interventions: Other: Nasal Secretion Sampling

INTERVENTIONS:
Other: Nasal Secretion Sampling — Nasal specimen collection will be performed at all visits. For every visit specimens will be collected using nasosorption FXi/PU (containing a synthetic absorptive matrix (SAM)), or a 10 cm-long plastic curette (nasosorption devices from Hunt Developments, UK) (Curette devices from Arlington Scientific, USA)

SUMMARY:
IgE-associated allergy is a hypersensitivity disease affecting more than 40% of the population in industrialised countries. Recently the kinetics of change of clinical and immunological parameters (e.g. nasal blockage and cytokine profiles) in response to allergen exposure have been described. Additionally through recent placebo controlled studies it has become clear that the response of certain cytokines can not only be triggered by allergen exposure but also mechanically e.g through the insertion of nasal swabs for collection of cytokines. However it is not clear to what extent the mechanically triggered cytokine responses may differ between healthy, allergic and asthmatic patients who have been shown to have different cytokine profiles in their nasal secretions and varying impairment of their respiratory epithelium. As collection devices for nasal secretions are frequently used in clinical studies, the investigators aim to assess the impact of mechanical stimulation by frequent cytokine sampling on the cytokine profile.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) and allergic asthma are a common manifestations of Type I allergy, an IgE-mediated hypersensitivity disease estimated to affect as much as 40% of the global population . IgE is produced by B cells and binds to the surface of mast cells and basophils via its high affinity Fce receptor I (FceRI). Crosslinking of surface IgE by its specific allergen induces degranulation of the cells as well as release of inflammatory mediators. This process which develops over minutes leads to the typical ocular, nasal and pulmonary symptoms of AR and asthma such as itching, reddening of the eyes, runny and/or congested nose and wheezing due to air trapping as a result of lower airway obstruction. Some patients may also develop late phase reactions (LPR). These responses typically develop 2-6 hours after allergen exposure, peaking in intensity between 6-9 hours and are mostly characterised by tissue oedema which manifests as airflow obstruction in the airways.

Since the introduction of easy to use and highly absorptive mucosal fluid sampling devices the mediators involved in the immediate and late phase allergic responses and the kinetics of their release have become well characterised over the past few years. Efforts by Imperial College London and unpublished data from the investigators group in Vienna have shown that key mediators involved in the immediate phase include mast cell derived mediators, (Tryptase, PGD2), epithelial alarmins (IL-33, sST2), and complement (C3a, C4a, C5a, D-Dimer). Mediators involved in the late phase reactions also include alarmins (sST2, TSLP), Th2 cytokines (IL-4, IL-5, IL-13), neutrophil mediators (MMP-9) and eosinophil mediators (EDN).

However what has also recently become clear through placebo controlled studies is that some mediators are mechanically mediated (unpublished observations), being released into the extracellular environment as a result of the sampling process itself. This is of vital interest as understanding which cytokines are mechanical and which are allergen specific will help guide future studies attempting to target specific biomarkers for treatment or disease monitoring. In order to understand if the mechanical release plays any role in the pathological response to allergens different patient cohorts will need to be investigated to see if their responses differ in any way.

Rational of the Study

In light of this the investigators propose a study to investigate the effects of mucosal sampling on cytokine release from nasal epithelium. The investigators plan to sample different patient cohorts (allergic rhinitis, allergic asthma, non-allergic) to see how mechanical effects are influenced by sampling and allergic or non-allergic status. By including 10 patients in each group the investigators hope to establish a range of "normal" for mechanical release of allergen relevant cytokines in each study group which will help inform future studies investigating allergen specific responses. In order to map both the symptomatic and objective responses to airway sampling, symptom scores and airway flow meters will be employed. To map the kinetics of responses the participants will undergo a mucosal sampling time course over the course of an 8 hour period on a single day. As no interventional substances are being given, this study will carry very low risk to the individuals involved while shedding important light on the epithelial responses to mechanical manipulation.

Study design In this single-center, pilot study a total of 36 patients (n=12 per group) will be recruited on a voluntary basis and will all receive nasal sampling. Study participants will undergo the nasal sampling in a single visit.

Screening Visit

Procedure:

* Signing of the Informed Consent Form
* Allocation of screening number
* Demographic Data
* History of allergy
* Assessment of In- and Exclusion Criteria
* Pregnancy test for females if requiring SPT
* Medical history
* Patients reporting a history of asthma will have to provide objective evidence of airway obstruction and reversibility (Spirometry reversibility or PC20 methacholine/histamine <8mg)
* Concomitant medication
* Anterior rhinoscopy
* Standard SPT with commercial extract from: hazel, ash, grass mix, ragweed, mugwort, D. pteronyssinus, D. farina, cat and dog dander, alternaria, cladosporium, histamine and negative control
* Blood sampling (max 60ml of heparinized blood and serum) - A part of the blood sample will be directly sent to the laboratory for analysis of total IgE, and specific IgE to relevant allergens. From the rest of the blood, RNA will be prepared and stored at -80°C and serum will be separated and stored at -20°C.
* nasal sampling (mucosal curette sampling and nasal secretion sampling)

Sampling Visit

Procedure:

* Reassessment of In and Exclusion Criteria (allergen-specific IgE results)
* Recording of concomitant medication
* Baseline Blood sampling
* Baseline nasal specimen collection for both nostrils (nasal secretion sampling) at 0min
* Baseline TNSS score
* Baseline PNIF
* Adverse event (AE) recording
* Blood, PNIF, nasal sampling (both nostrils: mucosal curette sampling and nasal secretion sampling), and TNSS score, 15min, 30min, 45min, 60min, 75min, 90min, 120min, 180min, 240min, 300min, 360min, 420min, 480min after onset of sampling timecourse

  4 Study procedures

4.1 Medical history of the participants, demographic data, concomitant medication The participants will be asked for their medical history including demographic data and concomitant medication, their allergic symptoms including intensity and duration and their allergic medication history.

4.2 History of allergy and TNSS score The participants will be asked for occurrence of sneezing, rhinorrhoea, nasal pruritus, nasal congestion and to grade each symptom. They will use the following symptom score method: 0 = absent; 1 = mild - present but easily tolerated; 2 = moderate - present, symptom is bothersome but not interfering with daily life activities; 3 = severe - symptom is difficult to tolerate and is interfering with daily life activities.

4.3 Anterior rhinoscopy Anterior rhinoscopy will be performed once during the screening visit to exclude anatomical variances (e.g. septal deviation) or pathological changes (e.g. nasal polyps). It will be performed by using a speculum with the patient seated with the head slightly back.

4.4 Peak Inspiratory Nasal Flow Meter (PNIF) The portability and ease of the PNIF provides a unique opportunity to obtain objective measurements. It has also recently been validated as a study tool during nasal allergen challenge.

4.4.1 Procedure: The PNIF uses a variable diameter tube calibrated directly in litres per minute along with a low inertia indicator ring. The position of the ring after an inspiratory manoeuvre indicates the maximum flow achieved. The device works when a patient inhales through the mouth or nose, this causes air to be drawn through the meter and a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale.

4.4.2 PNIF in study conduct: The participants will be trained how to use the PNIF on the day of the study and then it will be used at all study timepoints to gain information on nasal flow.

4.5 Skin prick test 4.5.1 Procedure: Allergens are inserted into the dermis of the forearm by gently pricking the skin through a drop (20ul) of an allergen-containing solution with a sterile lancet with at least 2 cm between each individual application point. 0.9% sodium chloride solution will be used as negative and histamine as positive control. In previously sensitized individuals, itchy swelling and a reddening of the skin (wheal and flare reaction) will occur within 15 minutes upon challenge with the respective allergen. After 20 minutes, allergen solutions will be wiped off and margins of the wheals will be traced with a ball point pen. Transparent tape will be bonded on the skin in order to transfer the outline of the wheal to the tape for the records. The surface of the wheals will be calculated by digital planimetry. For inclusion, wheals of at least 3 mm in diameter will be regarded as positive reactions.

4.5.2 Test solutions: A commercially available panel of tree and grass pollen, weed and perennial allergens (Allergopharma, Vienna, Austria) will be used at the screening visit and will be stored according to the manufacturer's instructions. As controls, sterile 0.9% NaCl solution (negative control) and histamine (positive control, Allergopharma, Vienna, Austria) will be used. They will be stored according to the manufacturer's instructions.

4.5.3 SPT in study conduct:

Screening Visit:

A standard skin prick test with commercial birch pollen extract and a panel of tree and grass pollen, weed and perennial allergens (all Allergopharma, Vienna, Austria) as used in routine diagnostic in the allergy clinic of the ENT department will be performed to assess the participants sensitization profile at the screening visit.

4.5.4 Safety precautions As a safety precaution, the participants will be monitored for 30 minutes after testing. All investigations will be done in the Outpatient Clinic of the ENT-Department, where full emergency equipment is available.

4.6 Blood sampling and measuring of immunological parameters Blood samples will be taken at the screening visit and at all study visits by puncture of the antecubital vein before skin testing. A maximum of 60ml per visit will be taken either heparinized (e.g. for basophil sensitivity assays) or for the preparation of serum (e.g. for assessment of total and allergen specific immunoglobulin levels or RBL assay). Serum vials will be processed and serum will be stored at -20°C. Allergen-specific IgE of blood samples of the screening visit will be measured by CAP-FEIA to assess the allergen-specific RAST-class of the patients. Measurement of total, free, and allergen-specific serum IgE, IgG, IgA and IgM will be performed either by CAP-FEIA, by microarray measurement or ELISA. Immune mediators will be measured using the MSD platform either by us or by our collaborators at AstraZeneca, Cambridge, UK. The measurement will be performed at the end of the study in all collected serum samples to minimize interassay variation.

4.7 Pregnancy testing In female participants, pregnancy will be excluded with a standard urine pregnancy test. The test will be performed before the first skin prick test at the screening visit and afterwards once a month.

4.8 Nasal specimen collection Nasal specimen collection will be performed at all visits. For every visit specimens will be collected using nasosorption FXi/PU (containing a synthetic absorptive matrix (SAM)), or a 10 cm-long plastic curette (nasosorption devices from Hunt Developments, UK) (Curette devices from Arlington Scientific, USA)

4.8.1 Nasosorption using FXi/PU (Hunt Developments, UK). Under visualization, the device will be inserted into the nasal cavity and be placed along the lateral wall against the inferior turbinate. The index finger of the patient will be used to press onto the external aspects of the alar and lateral nasal cartilages to hold the device in place. After 1 minute, the devices will be removed and then frozen at -80°C.

4.8.2 Mucosal mRNA sampling A 10cm nasal curette (either Rhino-Probe, Arlington Scientific, USA or Cellskim, Hunt Developments, UK) will be used. Under direct visualisation the curette will be brought to lie against the mid-inferior portion of the inferior turbinate. The curette will be pressed against the mucosal surface moved outwards 2-3 times. This motion will be repeated 2-3 times to ensure good sample collection. This curette and technique have been shown to cause no significant discomfort to participants and thus it has the advantage of no requirement for local anaesthetic. After collection Cells will be lysed in Qiagen RLT buffer and stored at -80°C for later mRNA analysis.

5 Investigational products and study medication 5.3 Concomitant medication 5.3.1 General All additional medication being taken by the subjects on entry to the study or at any time during the study are regarded as concomitant medication and will be documented in the CRF. Concomitant medications should be kept to a minimum during the study, but if considered necessary may be given if not interfering with the study protocol.

5.3.2 Rescue medication Although anaphylactic events are very unlikely in this study they always have to be considered possible. Therefore a complete emergency kit will be available immediately in case of anaphylactic reactions at SPT. Furthermore if the participant is suffering from strong skin symptoms after the SPT desloratadin 5mg will be provided to ameliorate the symptoms.

5.3.3 Prohibited concomitant medication

Subjects must remain off medications interfering with study procedures for the duration of the study. The following concomitant treatments are not permitted during this study:

* Systemic or topical corticosteroids
* Other immunosuppressant drugs
* Antihistamines or disodium cromoglycate 3 days prior to screening visit
* Systemic or intranasal adrenergic drugs
* Psychopharmacological drugs
* ACE-inhibitors or beta-blockers

  6 Adverse events An adverse event is any event during a clinical study, including intercurrent illness or accident, which impairs the well-being of the subject; it may also take the form of an abnormal laboratory value. The term adverse event does not imply a causal relationship with the study treatment.

All subjects experiencing adverse events - whether considered associated with the use of the study treatment or not - will be monitored until symptoms subside and any abnormal laboratory value has returned to baseline, or until there is a satisfactory explanation for the changes observed, or until death, in which case a full pathology report from a qualified pathologist will be provided. All findings must be reported on an "adverse event" page in the case record form.

All adverse events will be reported on and documented as described below. Adverse events are divided into the categories "serious" and "non-serious". This determines the procedure which must be used to report/document the adverse event (see below).

6.1 Definition of serious and non-serious adverse events

A serious adverse event is:

* Any event that is fatal or life-threatening
* Any event that is permanently disabling
* Any event that requires or prolongs hospitalization
* Any event that involves cancer, congenital abnormality, or occurs as a result of overdose (application of more than the stipulated dose).

Adverse events which do not fall into these categories are defined as non-serious.

6.2 Assessment of severity of AE

Regardless of the classification of an adverse event as serious or non-serious (see above), its severity must be assessed as mild, moderate or severe, according to medical criteria alone:

Mild = does not interfere with routine activities, acceptable Moderate = interferes with routine activities Severe = impossible to perform routine activities, considered as unacceptable by the physician, requires treatment, requires discontinuation of study, or has residual effect.

It should be noted that a severe adverse event need not be serious in nature. Regardless of severity, all serious adverse events must be reported on as below.

6.3 Reporting/documentation of adverse events Adverse events are collected by spontaneous reporting. 6.3.1 Reporting/documentation of serious adverse events All serious adverse events which occur during this study whether considered to be associated with the study or not, must be documented on an "Adverse event" page in the case record form.

A follow-up report including all new information obtained on the serious event must be prepared and will be collected.

The investigator will submit on request copies of all these reports to the ethics committee. Where necessary, investigators will inform the authorities.

6.3.2 Reporting/documentation of non-serious adverse events These are to be documented on an "Adverse event" page in the case record form.

7 Statistical analysis These analyses will seek to explore any statistically significant differences in longitudinal nasal cytokine trajectories between healthy individuals, atopic individuals and asthmatics. We will first undertake-basic descriptive statistics. Subject characteristics (e.g. health status, demographic variables) and outcome variables (e.g. nasal cytokine release, clinical responses) will be described by calculating maximum, minimum, median, mean and standard deviation for metric variables and absolute and relative frequencies for categorical variables for each subject group (healthy individuals, atopic individuals and asthmatics).

Log-changes from baseline will be compared between groups, and at each time point using t-tests for each pairwise comparison between groups, to explore the shape-of-trajectories-over-time. For graphical illustration, the individual log-baseline-change-trajectories of each patient will be plotted as well as group means with 95% CIs.

If log-changes-from-baseline-exhibit reasonable-linearity, we will test for an association between subject groups and longitudinal trajectories using mixed linear models with subject-specific random intercepts to account for intra-individual correlations of repeated measures, and group by time-interaction terms to test for statistically significant differences in trajectories. The motivation of this mixed modelling approach will be to increase-power-by-combining information-across multiple-time-points. Mean trajectories and 95% CIs as inferred by the mixed modelling work will also be plotted

8 Ethical and legal aspects The study will be carried out in keeping with local legal requirements and GCP. It will be performed in accordance with the guidelines of the Declaration of Helsinki (1964), including current revisions.

8.1 Informed consent of subject Before being admitted to the study, the subject must have consented to participate after the nature, scope and possible consequences of the clinical study have been explained in a form understandable to him/her. The subject must give consent in writing. The signature of the investigator will confirm the subject's consent. The patient may withdraw the consent, even without giving comments, at any time and without negative consequences for his future medical care. Nasosorption and/or RNA and/or blood samples may be sent in an anonymized form to collaboration partners outside Austria for analysis (e.g. analysis of cleaved and whole IL-33 by AstraZeneca, Cambridge UK). The patient is informed about this in the informed consent form.

8.2 Acknowledgement/approval of the study Before the start of the study, the study protocol will be submitted to the Ethics committee of the medical university Vienna and the general hospital of Vienna (Borschkegasse 8b/E 06, 1090 Vienna, Austria).

8.3 Insurance All subjects participating in this study will be insured at the Zürich Insurance company (Zürich-Versicherungs-Aktiengesellschaft, Schwarzenbergplatz 15, 1010 Vienna, Tel. +43 50 1255 1255).

8.4 Confidentiality All subjects' names will be kept secret in the investigators files. Subjects will be identified throughout documentation and evaluation by the number allotted to them during the study. The subjects will be told that all study findings will be stored and handled in strictest confidence.

9 Documentation and use of study findings 9.1 Documentation of study findings All results collected during the study will be collected in a source data file and will later be transferred to the case report forms (CRFs). All entries on the case record forms will be made legibly in black or blue ink. If corrections are made to entries in the case record form, the words or figures will be ringed and a single stroke drawn through them. The correct value will be entered beside the old entry and date and the correction will be initialled. Incorrect entries must not be covered with correcting fluid or obliterated or made illegible in any way. The completed CRFs will be signed by the investigator. CRFs will be completed immediately after the final examination. The medical records upon which the CRF is based will be kept for at least 15 years.

9.2 Use of the study findings The findings of this study will be published by the investigators in a scientific journal and presented in scientific meetings. The manuscript will be circulated to all co-investigators before submission.

10 Considerations on Potential Risks and Benefits for Study Participants and selection of dose

The included participants will not benefit directly from the study. However as the kinetics of mechanical mucosal stimulation is still not completely understood this comprehensive pilot study will provide an opportunity to guide future research which will hopefully lead to the discovery of novel therapeutic targets.

Potential risks for the participants include pain, infection and hematoma at the site of blood draw. During nasal mucosa and secretion sampling light nasal bleeding is a possible risk. During SPT, although highly unlikely, anaphylactic reactions are a possibility. To minimize risk of anaphylactic reactions and to provide optimal treatment in case an anaphylactic reaction should occur, patients will be monitored for a minimum of 30 minutes after SPT. At all participant visits trained personnel and emergency medication will be available all the time.

ELIGIBILITY:
Inclusion Criteria:

All groups

* Male or female
* 18 to 50 years of age
* Willingness to comply with the study protocol and written informed consent
* Subjects must have a standard health care insurance
* Subjects must be available during the study period to complete all treatments and assessments

Allergic Rhinitis

* Moderate to severe allergic rhinitis to grass pollen for at least two seasons according to medical history
* Skin prick test positive to grass pollen extract
* Blood ImmunoCAP sensitisation to grass pollen (>0.35 kU/L grass pollen extract specific IgE or higher as determined by UniCAP-FEIA)
* No history of Asthma

Allergic Asthma

* Clinical history of asthma
* Spirometry reversibility or PC20 methacholine/histamine <8mg
* Skin prick test positive to grass extract
* Blood ImmunoCAP sensitisation to grass pollen (>0.35 kU/L grass pollen extract specific IgE or higher as determined by UniCAP-FEIA)

Non-Allergics

* No history of Asthma
* No history of allergy
* Negative skin prick test to a common skin prick test panel including grass pollen
* No ImmunoCAP sensitisation to to grass pollen (<0.35 kU/L grass pollen extract specific IgE or higher as determined by UniCAP-FEIA)

Exclusion Criteria:

* Older than 50 or younger than 18 years
* Active smoker
* History of anaphylaxis
* Any severe chronic, malignant or general disease
* Treatment with systemic or topical (intranasal, inhaled, external) corticosteroids within the previous 2 months before the start of the study
* Treatment with antihistamines 3 days prior to the screening visit of the study
* Treatment with other immunosuppressant drugs within the previous 6 months prior to the start of the study
* Arterial hypertension or use of anti-hypertensive therapy, including beta-blockers
* Contra-indications to skin prick testing such as: skin inflammation in the test area, urticaria facticia
* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* Participation in another clinical trial within one month prior to the study; however participation during the previous month solely in the form of blood donation and/or without other interventions will be accepted
* Known alcohol or drug addiction or abuse
* Risk of non-compliance with the study procedure
* Previous immunotherapy with grass pollen
* Nasal polyps, history of chronic sinusitis or substantial deviation of the nasal septum

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Nasal cytokine responses to repeated mechanical stimulation in allergics, non allergics and asthmatics. | 1 Year
  The change in concentrations over time of a panel of relevant cytokines in Th2 immune responses e.g. IL-4, 5, 13 (all in pg/ml) will be measured using MSD multiplex assays to map responses to mechanical stimulation of the nasal mucosa.

SECONDARY OUTCOMES:
Changes in nasal airflow as a result of repeated nasal sampling | 1 Year
  The validated peak nasal inspiratory flow meter (PNIF) will be used to measure changes in nasal flow after nasal mucosa sampling.
Changes in nasal symptoms using the a validated nasal symptom scoring system | 1 Year
  In order to measure subjective changes in nasal symptoms after nasal mucosa sampling the total nasal symptom score (TNSS) will be used which contains the four parameters; nasal itch, nasal obstruction, sneezing and runny nose. Each parameter is scored from 0-3 with a higher score indicating a higher nasal symptom burden. The scores of each parameter are then added together to give the TNSS of which the maximum score is 12 and the lowest score is 0.
Defining differences in baseline and post sampling cytokine nasal mRNA levels | 1 Year
  Nasal tissue samples will be obtained using the validated Rhinoprobe device. The tissue samples with then be processed into RNA in order to measure any changes in cytokine mRNA levels before and after nasal sampling as a proxy to look for changes in gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schneider, MD, Principal Investigator — Attending ENT Specialist
Locations (1):
- 8H1.02, ENT Lab, Department of Otorhinolaryngology, Vienna General Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinberg EG. The Wao White Book on Allergy 2011-2012. Curr Allergy Clin Im. 2011;24(3):156-7.
- [Background] Bischoff SC. Role of mast cells in allergic and non-allergic immune responses: comparison of human and murine data. Nat Rev Immunol. 2007 Feb;7(2):93-104. doi: 10.1038/nri2018. PMID 17259966
- [Background] Valent P, Bettelheim P. The human basophil. Crit Rev Oncol Hematol. 1990;10(4):327-52. doi: 10.1016/1040-8428(90)90009-h. No abstract available. PMID 2278641
- [Background] Galli SJ, Tsai M, Piliponsky AM. The development of allergic inflammation. Nature. 2008 Jul 24;454(7203):445-54. doi: 10.1038/nature07204. PMID 18650915
- [Background] Leaker BR, Malkov VA, Mogg R, Ruddy MK, Nicholson GC, Tan AJ, Tribouley C, Chen G, De Lepeleire I, Calder NA, Chung H, Lavender P, Carayannopoulos LN, Hansel TT. The nasal mucosal late allergic reaction to grass pollen involves type 2 inflammation (IL-5 and IL-13), the inflammasome (IL-1beta), and complement. Mucosal Immunol. 2017 Mar;10(2):408-420. doi: 10.1038/mi.2016.74. Epub 2016 Sep 28. PMID 27677865
- [Background] Thwaites RS, Gunawardana NC, Broich V, Mann EH, Ahnstrom J, Campbell GA, Lindsley S, Singh N, Tunstall T, Lane DA, Openshaw PJ, Hawrylowicz CM, Hansel TT. Biphasic activation of complement and fibrinolysis during the human nasal allergic response. J Allergy Clin Immunol. 2018 May;141(5):1892-1895.e6. doi: 10.1016/j.jaci.2018.01.022. Epub 2018 Feb 7. No abstract available. PMID 29427640
- [Background] Downie SR, Andersson M, Rimmer J, Leuppi JD, Xuan W, Akerlund A, Peat JK, Salome CM. Symptoms of persistent allergic rhinitis during a full calendar year in house dust mite-sensitive subjects. Allergy. 2004 Apr;59(4):406-14. doi: 10.1111/j.1398-9995.2003.00420.x. PMID 15005764
- [Background] Boelke G, Berger U, Bergmann KC, Bindslev-Jensen C, Bousquet J, Gildemeister J, Jutel M, Pfaar O, Sehlinger T, Zuberbier T. Peak nasal inspiratory flow as outcome for provocation studies in allergen exposure chambers: a GA2LEN study. Clin Transl Allergy. 2017 Sep 17;7:33. doi: 10.1186/s13601-017-0169-4. eCollection 2017. PMID 28932387